CLINICAL TRIAL: NCT02165969
Title: Olfactory Function Following Endoscopic Endonasal Skull Base Surgery: Clinical and Histological Outcomes
Brief Title: Olfactory Function Following Endoscopic Endonasal Skull Base Surgery
Acronym: UPSIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ricardo L. Carrau, MD (Other)
Responsible Party: Sponsor-Investigator, Ricardo L. Carrau, MD, Professor, Ohio State University
Organization: Ohio State University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014H0063
Record Dates: First submitted 2014-05-23; First posted 2014-06-18 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Skull Base Pathology
Keywords: tumor; inflammatory process; fracture; defect
MeSH Terms: conditions — Neoplasms; Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- endoscopic endonasal surgery with UPSIT (Experimental): endoscopic endonasal surgery with UPSIT prior to surgery and at months 1, 3, 6, and 12 after surgery.
  Interventions: Procedure: endoscopic endonasal surgery with UPSIT

INTERVENTIONS:
Procedure: endoscopic endonasal surgery with UPSIT

SUMMARY:
The purpose of this study is to compare a subject's sense of smell before and after endoscopic endonasal surgery to remove a skull base abnormality (i.e. tumor, inflammatory process, fracture, defect, etc.) and use the information collected to validate approaches to surgery that will minimize side effects to the sense of smell function. Data will be collected using a smell identification test along with two questionnaires. In addition, demographic, medical history, treatment, outcome, and follow-up information will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with skull base pathologies requiring endonasal surgery at The Ohio State University Wexner Medical Center
* 18 years or older
* Able to consent for self
* Negative serum pregnancy test for women of childbearing potential

Exclusion Criteria:

* Patient unable to return to clinic at specific follow-up times
* Pregnant or nursing
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2014-06; Primary Completion 2017-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients with decreased olfactory function after endoscopic endonasal surgery | up to 12 months post surgery
  The subject will complete 2 questionnaires and the University of Pennsylvania Smell Identification Test (UPSIT) at baseline (pre-surgery) and at 1, 3, 6, and 12, months post surgery to determine if the sense of smell has been altered from surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Carrau, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States